CLINICAL TRIAL: NCT03687671
Title: Long-term Effects on Socioemotional Skills of Animal-assisted Therapy in Patients With Acquired Brain Injury
Brief Title: Long-term Effects of AAT in Patients With ABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Rehab Basel (Other); University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-01030
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries | interventions — Animal Assisted Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal-assisted therapy (Experimental): The intervention is animal-assisted occupational therapy, animal-assisted physiotherapy or animal assisted speech therapy with different animals. All animals are trained for the specific service with vulnerable patients. There are guinea pigs, rabbits, miniature pigs, sheeps, goats, chicken, dogs, cats and horses.
  Interventions: Other: Animal-assisted therapy
- Treatment as usual (activation program) (Active Comparator): As control intervention patients receive treatment as usual (TAU) in speech therapy, occupational therapy or physiotherapy. The control intervention is named activation program.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Animal-assisted therapy — Animal-assisted occupational therapy, animal-assisted physiotherapy and animal assisted speech therapy with different animals. All animals are trained for the specific service with vulnerable patients. There are guinea pigs, rabbits, miniature pigs, sheeps, goats, chicken, dogs, cats and horses.
  Arms: Animal-assisted therapy
Other: Treatment as usual — Speech therapy, occupational therapy or physiotherapy
  Other Names: activation program
  Arms: Treatment as usual (activation program)

SUMMARY:
The aim of this study is to investigate weather patients treated with animal-assisted therapy show better socioemotional skills compared to treatment as usual.

70 patients will be allocated randomly to one of two groups (control group and intervention group). During 6 weeks, all patients get two therapy sessions (AAT vs. TAU) per week. The 35 patients in the control group will get treatment as usual (TAU) in speech therapy, occupational therapy or physiotherapy twice a week whereas the 35 patients in the intervention group will get the same therapies but there will be an animal included in the therapy sessions.

The main outcome is the amount of expressed emotion and interaction in a standardized social situation measured via behavioral video coding.

Measurements will be done before the first therapy session (pre-measurement, t0) and after the last therapy session (post-measurement, t1) of the 6 weeks of intervention. The follow-up measurement will be done 6 weeks (follow-up I, t2) and 12 weeks later (follow-up II, t3).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented signed by the patient or his/her legal representative
* Inpatients of REHAB Basel with acquired brain injury and FIM-score over 60 (Funktionale Selbstständigkeitsmessung, Internationale Vereinigung für Assessment in der Rehabilitation, 1997)
* Minimum age of 18 years

Exclusion Criteria:

* Enrolment of the investigator, his/her family members, employees and other dependent persons
* medical contraindications for contact with animals as allergy, phobia etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
socioemotional behaviour | 18 weeks
  The amount of expressed emotion andsocial interaction in a standardized social situation measured via behavioral video coding.

SECONDARY OUTCOMES:
Social cognition | 18 weeks
  Measured via the "Movie for the Assessment of Social Cognition" MASC, Movie for the assessment of social cognition
  The MASC is a video based test, where 46 questions need to be answered. Correct answer = 1 point, incorrect answer = 0 point. The more questions are answered correctly the merrier the results are.
  Each question has four answer options. Each option has its own signification:
  a) correct ToM, b) exceeding ToM, c) less ToM, d) no ToM
  1. Emotion: 17 items, total score range 0-17
  2. Intention: 18 items, total score range 0-18
  3. Thoughts: 7 items, total score range 0-7
  Overall score range 0-46. The higher the score, the higher the capability of theory of mind (ToM).
  There is a rage of 30-39 right answered questions in healthy populations.
Therapy motivation | 18 weeks
  Measured with the questionnaire FPTM
  FPTM: Fragebogen zur Erfassung der Psychotherapiemotivation.
  Questionnaire measuring psychotherapy motivation with 39 items and 6 subscales:
  1. Physiological strain (Psychischer Ledensdruck): 10 itmens, total score range 10-40
  2. Hope for improvement (Hoffnung): 7 items, total score range 7-28
  3. Refuse of psychological need (Verneinung psychischer Hilfsbedürftigkeit): 7 items, score range 7-28
  4. Knowledge about treatment (Wissen): 5 items, total score range 5-20
  5. Initiative for treatment (Initiative): 4 items, total score range 4-16
  6. Symptom based care through others (Symptombezogene Zuwendung durch andere): 6 itmens, sore range 6-36
  Each question needs to be ranged from 1 to 4, high number mean higher motivation:
  1. = don't agree at all
  2. = don't agree
  3. = agree
  4. = totally agree
  Overall score range 39-156.
Quality of life score | 18 weeks
  Measured via the WHOQL-BREF
  WHOQL_BREF, World Health Organization Quality of Life
  Questionnaire about quality of life with 26 questions and four subscales:
  1. Physical health (Physische Gesundheit): 7 items, total score range 7-35
  2. Psychological health (Psychologische Gesundheit): 6 items, total score range 6-30
  3. Social relationship (Soziale Beziheungen): 3 items, total score range 3-15
  4. Environment (Umwelt): 8 items, total score range 8-40
  Each question needs to be ranged from 1 to 5, high number mean higher quality of life.
  1. = don't agree at all
  2. = don't agree
  3. = neutral
  4. = agree
  5. = totally agree
  Overall score range 26-130.
Depression | 18 weeks
  Measured via the BDI-FS
  BDI-FS, Beck Depressions-Inventar Fast Screening Questionnaire with 7 questions about negative feelings who need to be ranged from 0-3. High number mean higher rates in depression.
  0 = don't agree
  1. = agree little
  2. = agree
  3. = totally agree
  Overall score range 0-21.
Adherence to treatnemt | 6 weeks
  Percentage of completed therapy sessions

CONTACTS AND LOCATIONS:
Locations (1):
- REHAB Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided